CLINICAL TRIAL: NCT06930326
Title: A Prospective, Randomized, Triple-blind Comparative Study of Exosome and Exosomes-containing Formulation Versus Placebo in Treating Alopecia
Brief Title: Exosome Treatment and Hair Growth
Acronym: exosome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: COSMEDICIAN AP SDN BHD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UCSI-IEC-2022-FMHS-062.
Record Dates: First submitted 2025-03-24; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Alopecia Androgenica
Keywords: Alopecia
MeSH Terms: conditions — Alopecia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Group A), which received 0.9% sodium chloride (Placebo Comparator)
  Interventions: Other: 0.9 % NaCl
- Intervention group (Group B), received an Exosome-Containing Plant Extract Formulation (Experimental)
  Interventions: Other: intradermal exosome

INTERVENTIONS:
Other: intradermal exosome — The solution was drawn into five 1 mL tuberculin syringes, each fitted to a 30-gauge short needle. Intradermal injections of 0.05 to 0.1 mL per site were administered at approximately 1 cm apart, delivering a total volume of 5 mL per session.
  Arms: Intervention group (Group B), received an Exosome-Containing Plant Extract Formulation
Other: 0.9 % NaCl — The solution was drawn into five 1 mL tuberculin syringes, each fitted to a 30-gauge short needle. Intradermal injections of 0.05 to 0.1 mL per site were administered at approximately 1 cm apart, delivering a total volume of 5 mL per session.
  Arms: Control group (Group A), which received 0.9% sodium chloride

SUMMARY:
This study investigates a novel exosome-based plant formulation for treating male pattern baldness (androgenetic alopecia), a condition that affects self-esteem and well-being. Current treatments like minoxidil and finasteride offer limited effectiveness and may cause side effects, increasing demand for safer, more effective alternatives. Exosomes, small extracellular vesicles that facilitate cell repair and communication, show promise in promoting hair regeneration. Botanical extracts, such as Ecklonia cava (brown seaweed) and Thuja orientalis (medicinal plant), have also demonstrated hair growth benefits. This study combines these components into a single formulation to enhance therapeutic outcomes.

A randomized, double-blind, placebo-controlled trial is conducted to evaluate the efficacy of this exosome-containing formulation. The study enrolls 20 male participants aged 18 to 35 with Norwood 2-3 androgenetic alopecia. Participants are randomly assigned to receive either the exosome treatment (containing 10 billion exosomes with Ecklonia cava and Thuja orientalis extracts) or a placebo (0.9% sodium chloride). The treatment is administered through four biweekly sessions of intradermal scalp injections, performed by a certified aesthetic physician under strict aseptic conditions.

Hair growth is assessed using standardized photography, trichoscopic imaging, and hair density measurements, with a blinded medical assessor ensuring objective evaluation. Additionally, participants complete self-reported satisfaction surveys to gauge perceived effectiveness. Strict ethical guidelines are followed, including informed consent and exclusion of individuals with underlying medical conditions, recent hair treatments, or lifestyle factors that could influence results. The study aims to provide scientific evidence on the safety and efficacy of this exosome-based therapy as a potential alternative for hair restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Norwood grade 2-3 androgenic alopecia among male Malaysians.
2. Aged between 20 and 50 years.
3. Demonstrated the ability to comprehend the study protocol and information provided by the investigators.
4. Participants willing to give informed consent.

Exclusion Criteria:

1. Pre-existing thyroid disorders, bleeding disorders, or diabetes.
2. Current use of any medical hair treatment.
3. Corticosteroid or immunosuppressive drug use.
4. Alopecia classified as Norwood scale 1, 4, 5, 6, 7, or cicatricial alopecia.
5. Smoking.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Norwood grade 2-3 androgenic alopecia among male Malaysians.
Enrollment: 24 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Trichoscopic parameters: Total Hair Density | Baseline, 12, and 16 weeks post-treatment
  High-resolution trichoscopic images were captured using the Dino-Lite Trichoscope (Dino-Lite Europe, Almere, The Netherlands) at a standardized anatomical reference point, defined as the intersection of a vertical line descending from the lateral canthus of one eye (left or right) and a horizontal coronal line connecting both ears. Images were taken over two circular scalp areas, each with a diameter of 0.5 cm.
  These images were analyzed using Trichoscale Pro® software, which enables precise automated quantification of scalp structures. All measurements were subsequently verified manually by a blinded medical assessor to ensure accuracy.
  Total hair density was assessed as a primary parameter, with results expressed in hairs per square centimeter (hairs/cm²).
  The assessments were performed at baseline, 12, and 16 weeks post-treatment.
Modified global photographic assessment score (MGPA) | Baseline, 12 weeks, and 16 weeks post-treatment.
  Canon EOS 200D II digital camera (Canon, Taichung, Taiwan, China) was used for standardized profile photography, capturing lateral, facial, occipital, and cephalic views. The modified global photographic assessment score (MGPA) was used with the standardized 7-point rating score using scalp photographs: 1, significant disease progression; 2, moderate disease progression; 3, slight disease progression; 4, no change; 5, slight improvement; 6, moderate improvement; and 7, significant improvement. The scalp photographs of the subjects was evaluation of MGPA by blinded medical assessor. The assessments were performed at baseline, 12, and 16 weeks post-treatment.

SECONDARY OUTCOMES:
Hair Growth Satisfaction Scale (HGSS) | Baseline, and week 16
  Participants' self-perceived satisfaction with overall hair growth improvement will be evaluated using a Hair Growth Satisfaction Scale (HGSS) with Scale Range: 1 to 5.
  Scale Description:
  1. = Strongly Disagree
  2. = Disagree
  3. = Neutral
  4. = Agree
  5. = Strongly Agree Interpretation: Higher scores reflect greater participant satisfaction with hair growth results. A total satisfaction score (range: 5 to 25) will be computed by summing all item scores.
Trichoscopic parameters: Number of Empty Follicles | The assessments were performed at baseline, 12, and 16 weeks post-treatment.
  High-resolution trichoscopic images were obtained using the Dino-Lite Trichoscope (Dino-Lite Europe, Almere, The Netherlands) at a standardized anatomical reference point, defined as the intersection of a vertical line descending from the lateral canthus of one eye (either left or right) and a horizontal coronal line connecting both ears. Imaging was performed over two circular scalp areas, each with a diameter of 0.5 cm.
  The number of empty follicles was assessed. Image analysis was performed through manual verification by a blinded medical assessor to ensure accuracy. Results were expressed as the count of empty follicles per 0.5 cm circular area.
  The assessments were performed at baseline, 12, and 16 weeks post-treatment.
Trichoscopic Parameter: Percentage of Follicles with Peripilar Sign | The assessments were performed at baseline, 12, and 16 weeks post-treatment.
  High-resolution trichoscopic images were acquired using the Dino-Lite Trichoscope (Dino-Lite Europe, Almere, The Netherlands) at a standardized anatomical reference point, defined as the intersection of a vertical line extending from the lateral canthus of one eye (left or right) and a horizontal coronal line connecting both ears. Imaging was conducted over two circular scalp areas, each with a diameter of 0.5 cm.
  The percentage of follicles exhibiting the peripilar sign was evaluated. Visual scoring was performed on the trichoscopic images, with manual verification carried out by a blinded medical assessor to ensure measurement consistency. Results were reported as the proportion (%) of observed follicles displaying the peripilar sign.
  The assessments were performed at baseline, 12, and 16 weeks post-treatment.
Trichoscopic Parameter: Presence of Honeycomb Pigment Pattern (HCPP) | Assessments were conducted at baseline, 12 weeks, and 16 weeks post-treatment.
  High-resolution trichoscopic images were obtained using the Dino-Lite Trichoscope (Dino-Lite Europe, Almere, The Netherlands) at a standardized anatomical reference point, defined as the intersection of a vertical line extending from the lateral canthus of one eye (left or right) and a horizontal coronal line connecting both ears. Imaging was performed over two circular scalp areas, each with a diameter of 0.5 cm.
  The presence of the Honeycomb Pigment Pattern (HCPP) was assessed. Visual evaluation was conducted on the trichoscopic images by a blinded medical assessor to ensure consistency and objectivity. Results were reported in binary format as either present or absent.
  Assessments were conducted at baseline, 12 weeks, and 16 weeks post-treatment.
Trichoscopic Parameter: Presence of Fibrosis | Assessments were carried out at baseline, 12 weeks, and 16 weeks post-treatment.
  High-resolution trichoscopic images were captured using the Dino-Lite Trichoscope (Dino-Lite Europe, Almere, The Netherlands) at a standardized anatomical reference point, defined as the intersection of a vertical line extending from the lateral canthus of one eye (left or right) and a horizontal coronal line connecting both ears. Imaging was performed over two circular scalp areas, each with a diameter of 0.5 cm.
  The presence of follicular fibrosis was evaluated. Visual assessment was conducted using the trichoscopic images, with evaluations performed by a blinded medical assessor to ensure accuracy and minimize bias. Results were recorded in a binary format as either present or absent.
  Assessments were carried out at baseline, 12 weeks, and 16 weeks post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Dr. Edmond Ng Siah Chye, Principal Investigator — School of Healthy Ageing, Aesthetics & Regenerative Medicine, Faculty of Medicine and Health Sciences, UCSI University, Kuala Lumpur
Locations (1):
- Xeoul Clinic, Subang Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study are available from the corresponding authors on reasonable request. All of the individual participant data collected during the trial, after deidentification, will be shared upon reasonable request. Additional documents including study protocols, statistical analysis plans, informed consent forms, and clinical study reports will also be made available. The data will be available immediately following publication, with no end date. The data will be shared with anyone who wishes to access them on reasonable request. The data can be used for any type of analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available immediately following publication, with no end date. The data will be shared with anyone who wishes to access them on reasonable request.
Access Criteria: The datasets generated during and/or analyzed during the current study are available from the corresponding authors on reasonable request. All of the individual participant data collected during the trial, after deidentification, will be shared upon reasonable request. Additional documents including study protocols, statistical analysis plans, informed consent forms, and clinical study reports will also be made available. The data will be available immediately following publication, with no end date.